CLINICAL TRIAL: NCT02541669
Title: A Randomized, Open-Label and Double-Blind, Placebo-Controlled, Single- and Multiple-Dose, Phase 1 Study of the Pharmacokinetics of TAK-491 40 mg and 80 mg in Healthy Chinese Subjects
Brief Title: A Single- and Multiple-Dose Study of the Pharmacokinetics of TAK-491 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-491_112; U1111-1159-5559 (Other: WHO)
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer
Keywords: Drug therapy
MeSH Terms: interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- TAK-491 40 mg (Open Label) (Experimental): TAK-491 40 milligram (mg), tablet, orally, once daily on Day 1 and Days 4 to 10 as an open-label treatment.
  Interventions: Drug: TAK-491
- TAK-491 80 mg (Open-label) (Experimental): TAK-491 80 mg, tablet, orally, once daily on Day 1 and Days 4 to 10 as an open-label treatment.
  Interventions: Drug: TAK-491
- TAK-491 40 mg (Double-blind) (Experimental): TAK-491 40 mg, tablet, orally, once daily and TAK-491 80 mg placebo-matching tablet, orally, once daily on Day 1 and Days 4 to 10 in double-blind manner.
  Interventions: Drug: TAK-491; Drug: TAK-491 placebo
- TAK-491 80 mg (Double-blind) (Experimental): TAK-491 80 mg, tablet, orally, once daily and TAK-491 40 mg placebo-matching tablet, orally, once daily on Day 1 and Days 4 to 10 in double-blind manner.
  Interventions: Drug: TAK-491; Drug: TAK-491 placebo
- Placebo (Placebo Comparator): TAK-491 40 mg placebo-matching tablet, orally, once daily and TAK-491 80 mg placebo-matching tablet, orally, once daily on Day 1 and Days 4 to 10.
  Interventions: Drug: TAK-491 placebo

INTERVENTIONS:
Drug: TAK-491 — TAK-491 tablets
  Other Names: Azilsartan medoxomil; Edarbi
  Arms: TAK-491 40 mg (Double-blind); TAK-491 40 mg (Open Label); TAK-491 80 mg (Double-blind); TAK-491 80 mg (Open-label)
Drug: TAK-491 placebo — TAK-491 placebo-matching tablets
  Arms: Placebo; TAK-491 40 mg (Double-blind); TAK-491 80 mg (Double-blind)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of single- and multiple-dose of TAK-491 in healthy Chinese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-491. TAK-491 is being tested to treat people who have hypertension. This study will look at the pharmacokinetics of TAK-491 in Chinese participants who take TAK-491.

The study will enroll approximately 64 participants.

The first 16 enrolled participants have been randomly assigned (by chance, like flipping a coin) to 1 of the 2 treatment groups:

* TAK-491 40 mg
* TAK-491 80 mg

All participants will be asked to take 1 tablet at the same time on Day 1 and Day 4 to 10 during the study.

The following 48 randomized participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 3 treatment groups:

* TAK-491 40 mg
* TAK-491 80 mg
* TAK-491 placebo

All participants will be asked to take two tablets at the same time on Day 1 and Day 4 to 10 during the study.

This single-center trial will be conducted in China. The overall time to participate in this study is approximately 52 days. Participants will be admitted in the clinic for the first 12 days, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy adult male or female of Chinese descent.
4. Is aged 18 to 45 years, inclusive, at the time of informed consent and first study medication dose.
5. Has a body mass index (BMI) greater than or equal to (>=) 19.0 kilogram per square meter (kg/m^2) and less than (<) 24.0 kg/m^2, inclusive at Screening.
6. Has clinical laboratory evaluations (including clinical chemistry [fasted for at least 8 hours for the screening assessment], hematology, and complete urinalysis) within the reference range for the testing laboratory, unless the results were deemed by the investigator to be not clinically significant at Screening and Check-in (Day -1).
7. Is willing to refrain from strenuous exercise, from 72 hours before Check-in (Day-1) until after Final Visit.
8. A female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received TAK-491 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. Has history of uncontrolled, clinically significant manifestations of metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), endocrine, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, rheumatologic, skin and subcutaneous tissue disorders, infectious, hepatic, renal, urologic, immunologic, psychiatric or mood disorders (including any past history of suicide attempt), or a history of lactose intolerance, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of TAK-491 or other AII inhibitors or related compounds.
6. Has a positive urine drug result for drugs of abuse or breath alcohol test at Screening or Check-in (Day -1).
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Has taken any excluded medication, supplements, or food products.
9. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
10. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [example, cholecystectomy]).
11. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
12. Has positive test result for anti-Human immunodeficiency virus (HIV), anti- hepatitis C virus (HCV) antibodies, or for hepatitis B surface antigen (HBsAg) at Screening.
13. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).
14. Has poor peripheral venous access.
15. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
16. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participants with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
17. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than (>) 1.5 times the upper limits of normal.
18. Has a hemoglobin value <12 gram per deciliter (g/dL) at Screening.
19. Has a systolic blood pressure <110 and >=160 millimeter of Mercury (mmHg) or a diastolic blood pressure <60 and >=100 mmHg at Screening or Check-in (Day -1).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Beijing, Beijing,P.R., China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in China from 17 November 2015 to 17 March 2017.
Pre-assignment Details: Healthy Chinese participants were enrolled in the study in 2-parts, Open-label in which participants were allocated equally and randomly to TAK-491 40 milligram (mg) and TAK-491 80 mg and Double-blind in which participants were allocated equally and randomly to 1 of 3 regimens Placebo, TAK-491 40 mg, and TAK-491 80 mg.
Groups:
- Open Label: TAK-491 40 mg: TAK-491 40 mg, tablet, orally, once daily on Day 1 and Days 4 to 10 as an open-label treatment.
- Open Label: TAK-491 80 mg: TAK-491 80 mg, tablet, orally, once daily on Day 1 and Days 4 to 10 as an open-label treatment.
- Double-blind: Placebo: TAK-491 placebo-matching tablet, orally, once daily on Day 1 and Days 4 to 10 as a double blinded treatment.
- Double-blind: TAK-491 40 mg: TAK-491 40 mg, tablet, orally, once daily and TAK-491 placebo-matching tablets, orally, once daily on Day 1 and Days 4 to 10 as a double blinded treatment.
- Double-blind: TAK-491 80 mg: TAK-491 80 mg, tablet, orally, once daily and TAK-491 placebo-matching tablets, orally, once daily on Day 1 and Days 4 to 10 as a double blinded treatment.
Period: Open Label Treatment Period
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: Placebo | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Started | 8 | 8 | 0 | 0 | 0
Completed | 8 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Double-Blinded Treatment Period
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: Placebo | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Started | 0 | 0 | 16 | 16 | 16
Completed | 0 | 0 | 15 | 16 | 15
Not Completed | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: Placebo | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg | Total
Number analyzed (Participants) | 8 | 8 | 16 | 16 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The randomized set included all participants who were randomized.
  years | 28.8 (4.40) | 30.3 (4.98) | 33.0 (5.07) | 27.4 (4.19) | 29.7 (5.63) | 29.9 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The randomized set included all participants who were randomized.
  Participants
    Female | 3 | 3 | 1 | 1 | 3 | 11
    Male | 5 | 5 | 15 | 15 | 13 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The randomized set included all participants who were randomized.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 8 | 8 | 16 | 16 | 16 | 64
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: The randomized set included all participants who were randomized.
  participants
    China | 8 | 8 | 16 | 16 | 16 | 64
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The randomized set included all participants who were randomized.
  centimeter (cm) | 169.9 (6.66) | 165.3 (6.36) | 171.0 (6.07) | 170.4 (5.80) | 171.9 (6.75) | 170.2 (6.41)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The randomized set included all participants who were randomized.
  kilogram (kg) | 66.23 (4.785) | 59.83 (4.951) | 64.09 (6.012) | 64.79 (7.916) | 65.69 (6.934) | 64.40 (6.619)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The randomized set included all participants who were randomized.
  kilogram per square meter (kg/m^2) | 22.96 (1.289) | 21.94 (1.707) | 21.89 (1.143) | 22.23 (1.703) | 22.16 (1.109) | 22.18 (1.382)
Smoking classification [Count of Participants; unit: Participants] — Population: The randomized set included all participants who were randomized.
  Participants
    Never smoked | 8 | 8 | 14 | 14 | 13 | 57
    Current smoker | 0 | 0 | 0 | 0 | 0 | 0
    Ex-smoker | 0 | 0 | 2 | 2 | 3 | 7
Female Reproductive Status [Count of Participants; unit: Participants] — Population: The randomized set included all participants who were randomized.
  Participants
    Having Childbearing Potential | 3 | 3 | 1 | 1 | 3 | 11
    Postmenopausal | 0 | 0 | 0 | 0 | 0 | 0
    Surgically Sterile | 0 | 0 | 0 | 0 | 0 | 0
    Male Participants | 5 | 5 | 15 | 15 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536 (the Active Moiety Derived From TAK-491) on Day 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic (PK) set consisted of all participants who received study drug and had at least 1 measurable plasma concentration for TAK-536.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 16
nanogram per milliliter (ng/mL) | 2877 (25.0) | 6250 (20.5) | 2444 (22.5) | 5460 (30.4)

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536 (the Active Moiety Derived From TAK-491) on Day 10
Time Frame: Day 10 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: PK set where Day 10 assessments were available. The PK set consisted of all participants who received study drug and had at least 1 measurable plasma concentration for TAK-536.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 15
ng/mL | 3070 (4.6) | 6019 (29.5) | 2628 (23.3) | 6226 (19.9)

3. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-536 (the Active Moiety Derived From TAK-491) on Day 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK set consisted of all participants who received study drug and had at least 1 measurable plasma concentration for TAK-536.
Measure: Median (Full Range); unit: hour
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 16
hour | 3.03 [2.00 to 6.00] | 2.50 [2.00 to 4.00] | 3.00 [2.00 to 6.03] | 2.50 [1.00 to 6.00]

4. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-536 (the Active Moiety Derived From TAK-491) on Day 10
Time Frame: Day 10 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 15
hour | 3.00 [1.00 to 4.00] | 2.52 [2.00 to 6.00] | 3.49 [1.98 to 5.98] | 2.00 [1.98 to 6.00]

5. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-536 (the Active Moiety Derived From TAK-491) on Day 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 16
hour*nanogram per milliliter (h*ng/mL) | 25905 (27.3) | 50359 (12.1) | 23439 (22.6) | 45698 (32.1)

6. Primary Outcome: AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose for TAK-536 (the Active Moiety Derived From TAK-491) on Day 10
Time Frame: Day 10 pre-dose and at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 15
h*ng/mL | 25087 (21.5) | 45320 (14.7) | 21872 (19.1) | 47993 (31.8)

7. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for TAK-536 (the Active Moiety Derived From TAK-491) on Day 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
Number analyzed (Participants) | 8 | 8 | 16 | 16
hour | 11.18 (19.4) | 10.18 (24.1) | 11.12 (16.9) | 11.10 (18.9)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Day 40)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Open Label: TAK-491 40 mg | Open Label: TAK-491 80 mg | Double-blind: Placebo | Double-blind: TAK-491 40 mg | Double-blind: TAK-491 80 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8 | 6/16 | 4/16 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label: TAK-491 40 mg (N=8) | Open Label: TAK-491 80 mg (N=8) | Double-blind: Placebo (N=16) | Double-blind: TAK-491 40 mg (N=16) | Double-blind: TAK-491 80 mg (N=16)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 4
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1 | 3
Transaminases increased (Investigations) | 2 | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT02541669/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT02541669/SAP_001.pdf